CLINICAL TRIAL: NCT03602365
Title: Effects of Gentle Jogger on Oxygen Consumption
Brief Title: Gentle Jogger and Oxygen Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sackner Wellness Products LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GJHP2017COMP
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-09

CONDITIONS: Physical Inactivity; Oxygen Consumption
Keywords: Oxygen Consumption; Physical Activity; Passive Motion
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non randomized, single group study comparing the effects of GJ on resting oxygen consumption (VO2) measurements in seated and supine postures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OXYGEN CONSUMPTION SINGLE ARM (Experimental): Single arm Study Volunteer will h lie in supine posture for 20 min and oxygen consumption(VO2) will be measured in duplicate. Gentle Jogger (GJ) will be started in supine posture for 20 min and VO2 measured again in duplicate. The subject will be asked to sit in a chair for 20 min and VO2 will be measured in duplicate. Gentle Jogger (GJ) will be started in seated posture for 20 min and VO2 measured again in duplicate.
  Interventions: Device: Gentle Jogger (GJ)

INTERVENTIONS:
Device: Gentle Jogger (GJ) — Gentle jogger is a passive jogging device which passively moves the feet up and down simulating jogging

SUMMARY:
This is a non randomized study to determine the effects of Gentle Jogger(GJ), a passive jogging device on oxygen consumption in 2 postures supine and seated. Oxygen consumption measurements will be performed via indirect calorimetry in duplicate at rest ( supine and seated posture) , and repeated in duplicate during GJ (in supine and seated posture)

DETAILED DESCRIPTION:
The Gentle Jogger (GJ) is a patented non-FDA regulated wellness device in which GJ; 1) as part of a healthy lifestyle may help prevent certain chronic diseases or conditions such as heart disease, high blood pressure, and type 2 diabetes and 2) may help living well with certain chronic diseases or conditions such as heart disease, high blood pressure and type 2 diabetes. GJ is a passive simulated jogging device which moves the feet up and down passively, simulating jogging. GJ addresses the major health problem of physical inactivity.

This is a non randomized study of adult subjects on the effects of Gentle Jogger (GJ) on resting oxygen consumption (VO2).

This study will determine whether or not the use of GJ in either sitting or supine postures changes resting oxygen consumption, measured using indirect calorimetry method.

Potential study subjects will be invited to participate, and informed consent obtained from each subject.

Each subject will me asked to lie in supine posture for 20 mins followed by duplicate measurements of VO2. The GJ will be started in supine posture for 20 min followed by duplicate measurements of VO2. The subject will then be asked to sit in a chair for 20 min, followed by duplicate measurement of VO2, The GJ will be started for 20 min in seated posture followed by duplicate measurements of VO2.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects > 25 yrs old

Exclusion Criteria:

* Unable to provide informed consent
* Inability to follow command
* Physically unable to move feet up and down on a gentle jogger

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Change from Rest in Oxygen Consumption | After 20 min of Rest and after 20 min of Gentle Jogger
  oxygen consumption measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Sackner, MD, Study Director — CEO Sackner Wellness; Jose A Adams, MD, Principal Investigator — Director of Research Sackner Wellness
Locations (1):
- CIC Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sackner MA, Lopez JR, Banderas V, Adams JA. Can Physical Activity While Sedentary Produce Health Benefits? A Single-Arm Randomized Trial. Sports Med Open. 2020 Oct 2;6(1):47. doi: 10.1186/s40798-020-00278-3. PMID 33006749